CLINICAL TRIAL: NCT04834544
Title: A Randomized, Double-blind, Placebo-controlled, Preliminary Verifying Study About Safety and Efficacy of Maintenance DCVAC/OvCa After First-line Chemotherapy Added to Standard of Care in Patients With Newly Diagnosed FIGO III-IV Ovarian, Fallopian Tube, or Primary Peritoneal Carcinoma.
Brief Title: A Study of Maintenance DCVAC/OvCa After First-line Chemotherapy Added Standard of Care
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: SOTIO a.s. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IOV12
Record Dates: First submitted 2021-03-29; First posted 2021-04-08 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Epithelial Ovarian Carcinoma; Fallopian Tube Carcinoma; Primary Peritoneal Carcinoma
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DCVAC/OvCa arm (Experimental)
  Interventions: Combination Product: DCVAC/OvCa
- Placebo arm (Placebo Comparator)
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: DCVAC/OvCa — An active cellular immunotherapy product containing autologous dendritic cells that are generated ex vivo from patient's monocytes and apoptotic tumor cells prepared from tumor cell lines
  Arms: DCVAC/OvCa arm
Combination Product: Placebo — Placebo
  Arms: Placebo arm

SUMMARY:
This is a randomized, double-blind, placebo-controlled,parallel-group preliminary verifying study about safety and efficacy of maintenance DCVAC/OvCa after first-line chemotherapy added to standard of care in patients with newly diagnosed FIGO III-IV ovarian, fallopian tube, or primary peritoneal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Eighteen years of age or older at the time written informed consent is obtained
2. Newly diagnosed, histologically confirmed FIGO stage III or IV EOC (high-grade serous or high-grade endometrioid)
3. After primary debulking surgery or after interval debulking surgery; residual disease after surgery with optimal resection as R0 or R1 (R0 is defined as no macroscopic residual disease, R1 is defined as macroscopic residual disease with a maximal diameter of <1 cm)
4. Known BRCA status; if BRCA mutation status not known, results of BRCA testing must be available before randomization
5. Laboratory criteria:

   5.1. White blood cells >4000/mm3 (4.0×109/L) 5.2. Neutrophil count >1500/mm3 (1.5×109/L) 5.3. Hemoglobin ≥8 g/dL (80 g/L) 5.4. Platelet count ≥100,000/mm3 (100×109/L) 5.5. Total bilirubin <2× upper limit of normal (ULN) (benign hereditary hyperbilirubinemias, e.g., Gilbert's syndrome, are permitted) 5.6. Serum alanine aminotransferase, aspartate aminotransferase, and creatinine <2×ULN 5.7. Blood urea nitrogen <2×ULN
6. Adequate coagulation parameters:

   6.1. Activated partial thromboplastin time ≤1.5×ULN 6.2. International normalized ratio ≤1.5
7. ECOG performance status 0-2
8. Patients of child-bearing potential and their partners who are sexually active must agree to the use of 2 highly effective forms of contraception from the patient's signing of the ICF until 6 months after the last/final dose of first-line Pt-based adjuvant chemotherapy or IMP, whichever occurs later:

   a. Condom with spermicide and one of the following:
   * Oral contraceptive or hormonal therapy (e.g., hormone implants)
   * Placement of an intra-uterine device (IUD)

   Acceptable non-hormonal birth control methods include:
   1. Total sexual abstinence from the patient's signing of the ICF until 6 months after the last/final dose of first-line Pt-based adjuvant chemotherapy or IMP, whichever occurs later
   2. Vasectomized sexual partner plus male condom with spermicide and participant assurance that partner received post-vasectomy confirmation of azoospermia
   3. Tubal occlusion plus male condom with spermicide
   4. IUD plus male condom with spermicide. Provided coils are copper-banded.

   Acceptable hormonal methods include:
   1. Etonogestrel implants (e.g., Implanon, Norplan) plus male condom with spermicide
   2. Normal and low dose combined oral pills plus male condom with spermicide
   3. Norelgestromin/ethinyl estradiol transdermal system plus male condom with spermicide
   4. Intravaginal device plus male condom with spermicide (e.g., ethinyl estradiol and etonogestrel)
   5. Cerazette (desogestrel) plus male condom with spermicide. Cerazette is currently the only highly efficacious progesterone-based pill.
9. Signed informed consent and ability to comprehend its content

Exclusion Criteria:

1. Non-epithelial ovarian carcinoma or mixed epithelial histology
2. Borderline tumors (tumors of low malignant potential)
3. First-line Pt-based adjuvant chemotherapy already started after surgery
4. Intention to treat with intraperitoneal chemotherapy
5. Previous or concurrent radiotherapy to the abdomen and pelvis
6. Major surgery (with the exception of debulking surgery) within 3 weeks before informed consent signature or patient has not recovered from any effects of any major surgery
7. Malignancy other than EOC, except malignancy that has been in complete remission for a minimum of 3 years and except carcinoma in situ of the cervix or non-melanoma skin carcinomas that have been definitively treated
8. Use of any immunotherapy in the past (e.g., anti-PD-1/PD-L1 or other immune checkpoint inhibitors, therapeutic vaccines, adoptive cell therapy, cytokines); in case of uncertainty, discuss with the medical monitor
9. Symptomatic uncontrolled brain or leptomeningeal metastases. A scan to confirm the absence of brain metastases is not required. Patients with spinal cord compression may be considered if they have received definitive treatment for this and evidence of clinically stable disease for 28 days.
10. Co-morbidities:

    10.1. HIV positive 10.2. Active hepatitis B (HBV) and/or C (HCV), active syphilis 10.3. Evidence of active bacterial, viral, or fungal infection requiring systemic treatment 10.4. Clinically significant cardiovascular disease including: 10.4.1. Symptomatic congestive heart failure 10.4.2. Unstable angina pectoris 10.4.3. Severe cardiac arrhythmia requiring medication 10.4.4. Uncontrolled hypertension 10.4.5. Myocardial infarction or ventricular arrhythmia or stroke within a 6-month period before inclusion, ejection fraction <40% or serious cardiac conduction system disorders, if a pacemaker is not present 10.5. Pericardial effusion of any CTCAE grade 10.6. Severe chronic obstructive pulmonary disease defined as grade C and D according to Global Initiative for Obstructive Lung Disease 10.7. Patients considered a poor medical risk due to other serious, uncontrolled medical disorders, non-malignant systemic diseases or active, uncontrolled infections 10.8. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study treatment, or is not in the best interest of the patient to participate 10.9. Active autoimmune disease requiring treatment 10.10. History of severe forms of primary immune deficiencies 10.11. History of anaphylaxis or other severe reactions following vaccination 10.12. Psychiatric or social conditions which, in the investigator's opinion, would prevent participation in the study
11. Known hypersensitivity to any constituent of IMP
12. Systemic immunosuppressive therapy for any reason (except inhaled / intranasal steroids and short-term systemic steroids <30 days duration and ≤10 mg prednisone-equivalent per day are allowed)
13. Participation in a clinical trial using experimental therapy within the last 4 weeks before informed consent signature
14. Pregnant or breast feeding, or expecting to conceive children within the projected duration of the study treatment
15. Refusal to sign informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-04-19 (Actual); Primary Completion 2024-10-20 (Estimated); Study Completion 2027-04-20 (Estimated)

PRIMARY OUTCOMES:
Progress Free Survival | From randomization to the earlier date of assessment of objective progression or death by any cause in the absence of progression, the follow up period is about 2 years.
  PFS defined as the time from randomization to the earlier date of assessment of objective progression or death by any cause in the absence of progression; progression will be assessed by the investigator per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China